CLINICAL TRIAL: NCT00541749
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Escalating Single- and Multiple-Dose Study of the Safety, Tolerability, and Pharmacokinetics of rhuMAb IFNalpha in Adults With Systemic Lupus Erythematosus
Brief Title: A Study of rhuMAb IFNalpha in Adults With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IFN3958g
Record Dates: First submitted 2007-10-07; First posted 2007-10-10 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — rontalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: rhuMAb IFNalpha — Intravenous repeating dose

SUMMARY:
This is a Phase I, randomized, placebo-controlled, double-blind, dose-escalation study of single and repeat doses of rhuMAb IFNalpha, administered through the SC or IV route, in adults with Systemic Lupus Erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* For patients with reproductive potential (males and females), use of a reliable means of contraception (e.g., hormonal contraceptive, patch, vaginal ring, intrauterine device, physical barrier) throughout their participation in the study
* Diagnosis of SLE according to current American College of Rheumatology (ACR) criteria
* Disease duration of ≥ 1 year (after first diagnosis by a physician)
* Current immunity to measles, mumps, rubella, and varicella, as evidenced by positive IgG titers at the time of screening
* Current vaccination against influenza unless contraindicated in the investigator's judgment
* Normal Pap smear within the applicable time interval recommended by current American Cancer Society guidelines

Exclusion Criteria:

* Presence of active lupus nephritis
* Presence of active central nervous system (CNS) disease requiring treatment with high-dose corticosteroids or immunosuppressive agents
* Presence of active vasculitis requiring treatment
* History of arterial or venous thromboses within 12 months of screening
* Moderate to severe anemia, thrombocytopenia, or neutropenia
* Any manifestation likely to require, in the investigator's judgment, treatment with high-dose corticosteroids or the addition of an immunosuppressive regimen during the course of the trial
* Pregnancy or lactation
* Lack of peripheral venous access
* History of alcohol or substance abuse within 6 months of screening
* History of severe allergic or anaphylactic reactions to antibodies or fusion proteins
* Evidence of significant uncontrolled concomitant diseases
* Significant laboratory or electrocardiogram (ECG) abnormalities
* Evidence of any clinically significant abnormality on a chest X-ray
* Severly impaired renal function
* Impaired hepatic function
* Poorly controlled diabetes
* Conditions other than SLE that could require treatment with corticosteroids
* History of malignancy except completely excised basal cell carcinoma
* Congenital immune deficiency
* Positive tests for antibodies to HIV, hepatitis B (HBS antigen, anti-HBC) or C
* Positive IgM antibody titers in the presence of negative IgG titers to Epstein-Barr virus (EBV) or cytomegalovirus (CMV)
* Frequent recurrence of herpes lesions
* Episode of shingles within one year of screening
* Positive screening test for latent mycobacterium tuberculosis infection
* History of severe systemic bacterial, fungal, viral, or parasitic infections within the year prior to screening
* Any current or recent signs or symptoms of infection
* Received antibiotics orally (PO) during the 30 days prior to screening or IV antibiotics during the 60 days prior to screening
* Received a live vaccine within the 30 days prior to screening
* Has been hospitalized within the 30 days prior to screening
* Received > 20 mg/day prednisone for > 3 days during the 30 days prior to screening
* Received azathioprine, methotrexate, mycophenolate mofetil, cyclosporine, tacrolimus, sirolimus, pulse dose corticosteroids, intravenous immunoglobulin (IVIG), or transfusions within 6 months prior to screening
* Received cyclophosphamide within 2 years prior to screening
* Received a monoclonal antibody during the 12 months prior to screening
* Previously received an investigational treatment directed against interferon alpha
* Received B-cell depleting therapy (e.g., anti-CD20, anti-CD22)
* Received investigational treatment during the 30 days prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-02

PRIMARY OUTCOMES:
The incidence and nature of laboratory abnormalities | Length of study
The incidence, nature, and severity of adverse events | Length of study

SECONDARY OUTCOMES:
The PK profile of rhuMAb IFNalpha | Length of study
The incidence of antibodies directed against rhuMAb IFNalpha | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Jorn Drappa, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] McBride JM, Jiang J, Abbas AR, Morimoto A, Li J, Maciuca R, Townsend M, Wallace DJ, Kennedy WP, Drappa J. Safety and pharmacodynamics of rontalizumab in patients with systemic lupus erythematosus: results of a phase I, placebo-controlled, double-blind, dose-escalation study. Arthritis Rheum. 2012 Nov;64(11):3666-76. doi: 10.1002/art.34632. PMID 22833362